CLINICAL TRIAL: NCT00394186
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover, Phase IIa Study to Evaluate Efficacy and Safety of the Beta-3-Adrenergic Receptor Agonist Solabegron in Subjects With Irritable Bowel Syndrome
Brief Title: A Study To Investigate GW427353 In Subjects With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: B3I105940
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: GW427353; b3-Adrenergic Receptor Agonist; Irritable Bowel Syndrome (IBS); efficacy; tolerability; pharmacokinetics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — solabegron

INTERVENTIONS:
Drug: GW427353
Drug: Placebo
  Other Names: GW427353

SUMMARY:
This study will test the hypothesis that GW427353, a beta-3 adrenergic agonist, will relieve IBS pain or discomfort and associated symptoms in IBS patients.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of IBS which meets the Rome II criteria, screening pain score to be > 1.5 (0= no pain, 4 = very severe pain)

Exclusion Criteria:

* Subjects not meeting the Rome II criteria for the diagnosis of IBS
* Subjects with no stool for 7 days during the screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08

PRIMARY OUTCOMES:
completion of questionnaires by the subject, determining the average adequate relief rate | during the last 4 weeks of the treatment periods (weeks 3 to 6 in period 1 and weeks 15-18 in period 2)

SECONDARY OUTCOMES:
Blood levels of GW427353 | Week 1, 13
Questionnaire | Weeks 1, 6, 12, 18, 24
ECG, vital signs, adverse events | each visit
clinical lab tests | Weeks 1, 6, 12, 18, 24

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (16):
- Australia (7):
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Caboolture, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Spring Hill, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Malvern, Victoria
- France (5):
  - GSK Investigational Site, Issoire
  - GSK Investigational Site, Les Sables-d'Olonne
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Saint-Quentin
  - GSK Investigational Site, Vitry-sur-Seine
- Germany (4):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Berlin, State of Berlin